CLINICAL TRIAL: NCT02720445
Title: Long-Term Nicotine Treatment of Mild Cognitive Impairment
Brief Title: Memory Improvement Through Nicotine Dosing (MIND) Study
Acronym: MIND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Vanderbilt University (Other); Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Principal Investigator, Paul S. Aisen, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATRI-002-NIC; R01AG047992 (NIH); 131918 (Other: Food and Drug Administration (FDA))
Record Dates: First submitted 2016-03-22; First posted 2016-03-25 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Alzheimer's Disease; Nicotine; Transdermal Patch
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotine Transdermal Patch (Experimental): 190 participants will wear nicotine transdermal patches during waking hours. Active dose will titrate up from 3.5mg to 21mg in the first 6 weeks of treatment, remain at 21mg for 22.5 months, and then taper down in the final month of treatment
  Interventions: Drug: Nicotine Transdermal Patch
- Placebo Patch (Placebo Comparator): 190 participants will wear matching placebo patches during waking hours.
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Nicotine Transdermal Patch — 21mg Nicotine transdermal patches worn during waking hours. Active dose will titrate up from 3.5mg to 21mg in the first 6 weeks of treatment, remain at 21mg for 22.5 months, and then taper down in the final month of treatment.
  Arms: Nicotine Transdermal Patch
Drug: Placebo Patch — Matching placebo patches worn during waking hours.
  Arms: Placebo Patch

SUMMARY:
The purpose of the study is to see if daily transdermal nicotine is able to produce a significant cognitive, clinical and functional improvement in participants with MCI. Neuronal nicotinic receptors have long been known to play a critical role in memory function in preclinical studies, with nicotine improving attention, learning, and memory function.

The study will enroll 380 participants for a 2 year period. Participants will be randomized (50:50) to either the transdermal nicotine, beginning at 7mg/day, and increasing to 21mg/day, or placebo skin patch.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have a subjective memory concern as reported by participant, study partner, or clinician
2. Abnormal memory function documented by scoring within the education adjusted ranges on the Logical Memory II subscale (Delayed Paragraph Recall) from the Wechsler Memory Scale - Revised:

   * less than or equal to 11 for 16 or more years of education
   * less than or equal to 9 for 8 - 15 years of education
   * less than or equal to 6 for 0 - 7 years of education
3. Mini-Mental State Exam score between 24 and 30, inclusive
4. Clinical Dementia Rating (CDR) Global = 0.5. Memory Box score must be at least 0.5
5. General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's disease dementia cannot be made by the site physician at the time of the screening visit
6. Age 55-90 (inclusive)
7. Stable permitted medications for 4 weeks or longer as specified in Section 6, including:

   • Memantine and cholinesterase inhibitors are allowable if stable for 12 weeks prior to screen
8. Geriatric Depression Scale score of less than or equal to 14
9. Study Partner is available who has frequent contact with the participant (e.g. an average of 10 hours per week or more), and can accompany the participant to most visits to answer questions about the participant
10. Adequate visual and auditory acuity to allow neuropsychological testing
11. Good general health with no additional diseases/disorders expected to interfere with the study
12. Participant is not pregnant, lactating, or of childbearing potential (i.e. women must be two years post-menopausal or surgically sterile)
13. Completed six grades of education or has a good work history
14. Fluent in English or Spanish

Exclusion Criteria:

1. Regular use of tobacco products within the past year, such as smoking (cigarettes, pipes, cigars, etc.) or use of other nicotine products (chewing tobacco, e-cigarettes, nicotine patches, gum, sprays, etc.).
2. Any significant neurologic disease such as Alzheimer's disease dementia, Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
3. Major depression, bipolar disorder as described in DSM-V within the past 1 year or psychotic features, agitation or behavioral problems within 3 months, which could lead to difficulty complying with the protocol
4. History of schizophrenia (DSM V criteria)
5. History of alcohol or substance abuse or dependence within the past 2 years (DSM V criteria)
6. Clinically significant or unstable medical condition, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic disease in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results, or the participant's ability to participate in the study.
7. Has had a history within the last 5 years of a primary or recurrent malignant disease with the exception of non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with normal prostate-specific antigen post-treatment
8. Clinically significant abnormalities in B12 or TFTs (Thyroid Function Tests) that might interfere with the study. A low B12 is exclusionary, unless the required follow-up labs (homocysteine (HC) and methylmalonic acid (MMA)) indicate that it is not physiologically significant.
9. Clinically significant abnormalities in screening laboratories or ECG.
10. Residence in skilled nursing facility.
11. Use of any excluded medication as described in the protocol, including:

    * Use of centrally acting anti-cholinergic drugs
    * Use of any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening.
12. For CSF sub-study participants, a current blood clotting or bleeding disorder, or significantly abnormal PT or PTT (partial thromboplastin time) at screening
13. For MRI sub-study participants, contraindications for MRI studies, including claustrophobia, the presence of metal (ferromagnetic) implants, or cardiac pacemaker.
14. Patients whom the Site PI deems to be otherwise ineligible.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Cogstate Battery International Shopping List Test - Total Immediate Recall (ISLT-TIR) | 2 years

SECONDARY OUTCOMES:
Change from Baseline in Mild Cognitive Impairment - Clinical Global Impression of Change (MCI-CGIC) to Month 25 | 2 years
  The MCI-CGIC is the MCI version of the clinician's global impression of change. In this trial it will measure change in the participant's condition between the baseline visit and subsequent visits.
Change from Baseline in Cogstate Brief Battery (CBB) to Month 25 | 2 years
  This battery will be used for the purpose of assessing the cognitive status of the participants and will assist in documenting multiple domains of cognitive impairment.
Change in Baseline in New York University (NYU) Paragraph Recall to Month 25 | 2 years
  This test measures immediate and delayed verbal recall of a brief story.
Change from Baseline in Clinical Dementia Rating Scale (CDR) - Sum of Boxes (SOB) to Month 25 | 2 years
  The is a clinical scale that rates the severity of dementia as absent, questionable, mild, moderate, or severe.
Change in Baseline in Geriatric Depression Scale (GDS) to Month 25 | 2 years
  This is a 30-item self-report assessment used to identify depression in the elderly.
Change in Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL) to Month 25 | 2 years
  This scale is an inventory developed to assess functional performance in participantss with Alzheimer's disease.
Change from Baseline in Older Adult Self Report (OASR) / Older Adult Behavior Checklist (OABCL) to Month 25 | 2 years
  The OASR/OABCL is a general index of psychopathologic symptoms and signs that is specifically relevant to elderly individuals and is developmentally appropriate, covers a wide range of psychopathologic signs and symptoms, and functional measures. It allows multi-informant perspective (both patient and informant). The items are focused on common elderly emotional, functional, or medical problems. The OASR is completed by the participant and the companion OABCL is completed by the informant.

OTHER OUTCOMES:
Change from Baseline in Cerebral Spinal Fluid (CSF) Biomarkers to Month 25 | 2 years
  CSF will be performed in approximately 50 participants each
Change from Baseline of Volumetric Magnetic Resonance Imaging (vMRI) to Month 25 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Aisen, MD, Study Director — USC Alzheimer's Therapeutic Research Institute (ATRI); Paul Newhouse, MD, Study Director — Vanderbilt University
Locations (36):
- United States (36):
  - Perseverance Research Center, Scottsdale, Arizona
  - Central Arkansas Veterans Healthcare System, North Little Rock, Arkansas
  - USC Rancho Los Amigos, Downey, California
  - Sharp Neurocognitive Research Center, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Nuvance Health Medical Practice Ct, Inc.; Associated Neurologists, PC, Danbury, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Brain Matters Research, Stuart, Florida
  - Augusta University Movement and Memory Disorders, Augusta, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Headlands Eastern MA LLC, Plymouth, Massachusetts
  - University at Buffalo (UBMD), Buffalo, New York
  - Velocity Clinical Research - Syracuse, East Syracuse, New York
  - New York University Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Integrative Clinical Trials, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Central States Research (formerly Tulsa Clinical Research), Tulsa, Oklahoma
  - Providence Brain and Spine Institute, Portland, Oregon
  - LeHigh Valley Hospital, Allentown, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Ralph H. Johnson VA Health Care System, Charleston, South Carolina
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Neurological Institute, Houston, Texas
  - Glenn Biggs Institute at the University of Texas Health, San Antonio, Texas
  - University of Washington Memory and Brain Wellness Center, Seattle, Washington
  - Kingfisher Cooperative, LLC, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Newhouse PA, Potter A, Corwin J, Lenox R. Age-related effects of the nicotinic antagonist mecamylamine on cognition and behavior. Neuropsychopharmacology. 1994 Apr;10(2):93-107. doi: 10.1038/npp.1994.11. PMID 8024677
- [Background] Newhouse P, Kellar K, Aisen P, White H, Wesnes K, Coderre E, Pfaff A, Wilkins H, Howard D, Levin ED. Nicotine treatment of mild cognitive impairment: a 6-month double-blind pilot clinical trial. Neurology. 2012 Jan 10;78(2):91-101. doi: 10.1212/WNL.0b013e31823efcbb. PMID 22232050
- [Background] Dumas J, Hancur-Bucci C, Naylor M, Sites C, Newhouse P. Estrogen treatment effects on anticholinergic-induced cognitive dysfunction in normal postmenopausal women. Neuropsychopharmacology. 2006 Sep;31(9):2065-78. doi: 10.1038/sj.npp.1301042. Epub 2006 Feb 15. PMID 16482084
- [Background] Newhouse PA, Dumas J, Hancur-Bucci C, Naylor M, Sites CK, Benkelfat C, Young SN. Estrogen administration negatively alters mood following monoaminergic depletion and psychosocial stress in postmenopausal women. Neuropsychopharmacology. 2008 Jun;33(7):1514-27. doi: 10.1038/sj.npp.1301530. Epub 2007 Aug 15. PMID 17700646
- [Background] Newhouse PA, Sunderland T, Tariot PN, Blumhardt CL, Weingartner H, Mellow A, Murphy DL. Intravenous nicotine in Alzheimer's disease: a pilot study. Psychopharmacology (Berl). 1988;95(2):171-5. doi: 10.1007/BF00174504. PMID 3137593
- [Derived] Joe E, Ringman JM. Cognitive symptoms of Alzheimer's disease: clinical management and prevention. BMJ. 2019 Dec 6;367:l6217. doi: 10.1136/bmj.l6217. PMID 31810978
- See also: Alzheimer's Therapeutic Research Institute (ATRI). ATRI is the Coordinating Center for the MIND study. — http://keck.usc.edu/atri/research/studies/
- See also: MIND study public website — http://mindstudy.org/